CLINICAL TRIAL: NCT06115408
Title: Evaluation of Using Dienogest and N-Acetyl Cysteine on the Volume of Uterine Leiomyoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Esraa Mosaad Awd El-sayed, Researcher,ob/gyn Resident, Principal Investigator, Esraa Awd, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Leiomyoma volume reduction
Record Dates: First submitted 2023-03-09; First posted 2023-11-03 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Uterine Leiomyoma
Keywords: Fibroids dienogest NAC
MeSH Terms: conditions — Myofibroma | interventions — dienogest; Acetylcysteine

STUDY DESIGN:
Intervention Model Description: The study will be conducted on 40 women; they will be subdivided into 2equal groups .each group receive different intervention
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug;Dienogest (Experimental): 2mg pills oral daily
  Interventions: Drug: Dienogest 2 MG
- Drug;N-Acetylcysteine (Experimental): 600 mg/day oral daily
  Interventions: Drug: N-acetyl cysteine

INTERVENTIONS:
Drug: Dienogest 2 MG — Clinical trial
  Other Names: Gynoprogest
  Arms: Drug;Dienogest
Drug: N-acetyl cysteine — Clinical trial
  Other Names: Gemacysteine
  Arms: Drug;N-Acetylcysteine

SUMMARY:
This 2 arm randomized clinical trial will assess the impact of Dienogest and N-Acetyl Cysteine on volume reduction of uterine leiomyoma

DETAILED DESCRIPTION:
Group A women will receive Dienogest orally 2mg pills daily for 3 months .20 cases Group B women will receive NAC orally at a dose of 600 mg/day for 3 months ,20 cases

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-45 years.
2. Women with uterine leiomyoma (sub-mucous, sub-serous or intramural) based on transvaginal sonography criteria. Uterine fibroids most often appear as concentric, solid, hypoechoic masses. This appearance results from the prevailing muscle, which is observed at histologic examination. These solid masses absorb sound waves and therefore cause a variable amount of acoustic shadowing.
3. Regular menstruation: regular period interval from 21 to 35 days.

Exclusion Criteria:

1. Pregnant or menopausal women.
2. History of malignancies, metabolic, hematologic, cardiac, thromboembolism, diabetes, renal or hepatic diseases.
3. History of hormonal drug use or treatment for leiomyoma in the past 3 months.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
leiomyoma size reduction | 3 months
  vertical x horizontal diameter in mm by transvaginal U/S

SECONDARY OUTCOMES:
Dysmenorrhea | 3 Monthes
  according to the visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain)
heavy menstrual bleeding | 3 months
  assess by PBAC score
blood loss | 3 months
  by hemoglobin level

CONTACTS AND LOCATIONS:
Overall Officials: Amr Mahmoud, lecturer, Study Chair — Ain Shams University; Ahmed mohamed mamdouh, assisstant professor, Study Chair — Ain Shams University
Locations (1):
- Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All of individual participant data collecting during the trial ,after deidentification
Supporting Information: Study Protocol
Time Frame: Immediately following publication.no end date
Access Criteria: Any purpose
URL: https://med.asu.edu.eg

DOCUMENTS (3):
  • Study Protocol (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT06115408/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT06115408/SAP_001.pdf
  • Informed Consent Form (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT06115408/ICF_002.pdf